CLINICAL TRIAL: NCT03390712
Title: Mirror-image Study Exploring Relapse and Resource Utilization of Paliperidone Palmitate and Risperidone Long-acting Injection in Vitalité Health Network Patients
Brief Title: Mirror-image Study of Paliperidone Palmitate and Risperidone Long-acting Injection
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Réseau de Santé Vitalité Health Network (Other)
Collaborators: Janssen Inc. (Industry)
Responsible Party: Principal Investigator, Michael Kemp, Psychiatric Pharmacist and Clinical Researcher, Réseau de Santé Vitalité Health Network
Other Study IDs: PHAR-1701
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: Paliperidone palmitate; Risperidone long-acting injection; mirror-image
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Paliperidone Palmitate; Risperidone; Antipsychotic Agents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paliperidone Palmitate: Patients who have received a minimum of 3 months of treatment with an injection of paliperidone palmitate.
  Interventions: Drug: Paliperidone Palmitate; Drug: Antipsychotic
- Risperidone Long-acting injection.: Patients who have received a minimum of 3 months of treatment with Risperidone long-acting injection.
  Interventions: Drug: Risperidal Consta; Drug: Antipsychotic

INTERVENTIONS:
Drug: Paliperidone Palmitate — Monthly injections
  Other Names: Invega Sustenna
  Groups: Paliperidone Palmitate
Drug: Risperidal Consta — Bi-weekly injection
  Other Names: Risperidone long-acting injection
  Groups: Risperidone Long-acting injection.
Drug: Antipsychotic — Any oral antipsychotic prescribed to be taken on a regular basis prior to the initiation of a long-acting injectable antipsychotic.
  Other Names: Oral antipsychotics

SUMMARY:
The primary objective of this single-center multi-site retrospective chart review is to determine if paliperidone palmitate and/or risperidone long-acting injection can decrease the number of psychiatric relapses following their initiation in an inpatient acute psychiatric unit compared to oral antipsychotic therapy and determine if one treatment is superior to the other in this regard. This study will utilize a mirror-image design and incorporate up to a 3 years of follow-up following the index admission. Secondary objectives of this study will be to determine the change in hospital resource utilization for psychiatric reasons following treatment initiation, and to determine the difference in time to relapse.

ELIGIBILITY:
Inclusion Criteria:

• Patients who were initiated on either Risperidone long-acting injection or Paliperidone palmitate during an acute psychiatric admission for schizophrenia or other psychotic related disorders.

Exclusion Criteria:

* Patients who had their long-acting injection stopped prior to the discharge date of their index admission.
* Patients who received a long-acting injection in the year prior to the index admission.
* Patients who had a psychiatric admission to a forensic, rehabilitation or high dependency unit during the observation period prior to or following their index admission.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients initiated on long-acting injectable anipsychotics from the regional hospitals under the direction of the Vitalité health network.
Sampling Method: Non-Probability Sample
Enrollment: 328 (Estimated)
Dates: Start 2018-01-02 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Psychiatric Relapse | up to 3 years
  Hospitalizations will be used as a proxy for relapse and the primary endpoint will be the number of hospital admissions following the discharge date of the index admission for up to 3 years compared to an equivalent timeframe prior to the beginning of the index admission (and including the 1st day of the index admission). Patients will be considered eligible for the primary objective after 3 months of continued long-acting injection treatment.

SECONDARY OUTCOMES:
Hospital Resource utilization for psychiatric reasons | up to 3 years
  Number of ER visits for psychiatric reasons, number of days admitted in hospital for psychiatric reasons.
Time to relapse | up to 3 years
  time following discharge of index admission until the subsequent admission for psychiatric reasons (in days); time following discharge of index admission until the subsequent ER visit for psychiatric reasons (in days).

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Chaleur Regional Hospital, Bathurst, New Brunswick
  - Campbellton Regional Hospital, Campbellton, New Brunswick
  - Edmundston Regional Hospital, Edmundston, New Brunswick
  - Dr. George-L.-Dumont University Hospital Center, Moncton, New Brunswick

IPD SHARING:
Plan to Share IPD: No